CLINICAL TRIAL: NCT00869986
Title: A Double Blind, Placebo Controlled Multi-Center Study to Evaluate the Efficacy and Safety of MBP8298 in Relapsing Remitting Multiple Sclerosis
Brief Title: A Study for Patients With Relapsing Remitting Multiple Sclerosis
Acronym: MINDSET01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: BioMS Technology Corp. (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12791; I3E-BM-MSAE; 2006-001947-70; MBP8298-RR01
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — MBP-8298

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dirucotide (Experimental)
  Interventions: Drug: dirucotide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dirucotide — 500mg, intravenous, every 6 months for 15 months
  Other Names: MBP8298; LY2820671
  Arms: Dirucotide
Drug: placebo — intravenous, once every six months for 15 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to test if dirucotide is safe and effective in treating patients with relapsing remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-50 years of age
2. Relapsing-remitting multiple sclerosis (RRMS) according to "Diagnostic criteria for multiple sclerosis: 2005 revisions to the McDonald Criteria" (Annals of Neurology 58: 840-846)
3. At least 2 years history of MS before trial entry
4. Documented history of 2 or more exacerbations in the 2 years prior to trial entry
5. Stable neurological status for at least 30 days before first study drug administration
6. Have an EDSS from 0-5.5
7. If female, she must either

   * be post-menopausal or surgically sterilized; or
   * use a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study; and
   * be neither pregnant nor breast-feeding
8. Willingness and ability to comply with the protocol for the duration of the study
9. In the Investigator's opinion, subjects must be reliable, compliant, and agree to cooperate with all trial evaluations
10. Subject must be able and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with regulatory requirements

Exclusion Criteria:

1. Have Clinically Isolated Syndrome (CIS), Secondary Progressive MS (SPMS), Primary Progressive MS (PPMS)
2. Any known malignancy, or history of malignancy, with the exclusion of basal cell carcinoma
3. Have active, clinically significant liver, renal or bone marrow disease accompanied with significant laboratory abnormalities in the range of grade I or more as defined by Common Toxicity Criteria (CTC),
4. Clinically significant ECG abnormalities at screening
5. Have the presence of systemic disease that, in the opinion of the investigator, might interfere with subject safety, compliance or evaluation of the condition under study (e.g. insulin dependent diabetes, lyme disease, clinically significant cardiac, hepatic, or renal disease, Human Immunodeficiency Virus, or Human T-Cell Lymphotrophic Virus Type-1)
6. Have current autoimmune disease, compromised immune function or infection
7. History of allergic reactions to glatiramer acetate
8. Steroid therapy within 30 days prior to first study specific procedure, or any other treatment known to be used for putative or experimental MS treatment
9. Therapy with ß-interferon, glatiramer acetate, statins, copaxone or nonspecific phosphodiesterase inhibitors within 3 months prior to first study-specific test
10. Therapy with mitoxantrone, cyclophosphamide, methotrexate, azathioprine, or any other immuno-modulating (e.g. IVIG) or immunosuppressive drugs including recombinant or non-recombinant cytokines or plasma exchange within 6 months prior to performance of the first study-specific test, with the exception of corticosteroids or ACTH for relapse treatment
11. Treatment at any time with an altered peptide ligand, cladribine, total lymphoid irradiation, monoclonal anti-body treatment e.g. anti-CD4, anti-CD52, anti-VLA4, Anti-CD20,
12. Any contraindications for MRI, e.g. pacemaker or known allergy to Gadolinium- DTPA
13. Participation in any other trial of an investigational agent within 90 days prior to screening
14. History of alcohol or drug abuse as specified by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) within the year before screening
15. Any medical, psychiatric or other condition that could result in a subject not being able to give fully informed consent, or to comply with the protocol requirements
16. Any other condition that, in the Investigator's opinion, makes the subject unsuitable for participation in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Annualized relapse rate | 15 months

SECONDARY OUTCOMES:
Time to confirmed worsening of disability by Expanded Disability Status Scale (EDSS) | baseline, 15, 24 and 27 months
Time to confirmed worsening of disability by Multiple Sclerosis Functional Composite (MSFC) | baseline, 15, 24 and 27 months
Proportion of patients relapse-free | 15, 24, and 27 months
Activity analysis of T2 and Gadolinium enhancing lesions | 15 and 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9am - 5pm Eastern Time (UTC/GMT)-5 hours,EST), Study Director — Eli Lilly and Company
Locations (6):
- Military Medical Academy, Sofia, Bulgaria
- Silesian Medical School, Katowice, Poland
- Clinical City Hospital No. 11, Moscow, Russia
- Clinical Center of Serbia, Belgrade, Serbia
- FNsP J A Reimana, Prešov, Slovakia
- Vinnitsa State Medical University, Vinnitsa, Ukraine